CLINICAL TRIAL: NCT00692874
Title: Quality of Life Analysis of Prostate Cancer Patient's Therapy
Brief Title: Quality of Life Analysis of Treatment in Patients With Prostate Cancer on Adjuvant Zoladex Therapy
Acronym: AZTEK EXT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar Medical Science Director, AstraZeneca
Other Study IDs: NIS-OHU-ZOL-2007/1
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Prostate Cancer
Keywords: Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open label, non-interventional quality of life analysis for Zoladex treated prostate cancer patients by investigator's questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Early or locally-advanced prostate cancer patients on androgen deprivation therapy
* Investigators are requested to recruit patients only with at least 1 month prior Zoladex treatment.

Exclusion Criteria:

* Allergy to substance of medication
* Prostate cancer patients with advanced disease

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Early or locally-advanced prostate cancer patients on androgen deprivation therapy
Sampling Method: Non-Probability Sample
Enrollment: 1646 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Elements of a general and three disease-specific investigator questionnaire | Quarterly (plus or minus 3 days )

SECONDARY OUTCOMES:
Investigator Assessment Report | Yearly (plus or minus 1 week )

CONTACTS AND LOCATIONS:
Overall Officials: Péter Tenke, M.D., Principal Investigator — "Jahn Ferenc" City Hospital Budapest; Csaba Csongvai, Study Director — AstraZeneca Hungary; Éva Gulyás, Study Chair — AstraZeneca Hungary
Locations (20):
- Hungary (20):
  - Research Site, Baja
  - Research Site, Békés
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Dunaújváros
  - Research Site, Érd
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kiskunhalas
  - Research Site, Nagykőrös
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szentendre
  - Research Site, Székesfehérvár
  - Research Site, Tatabánya
  - Research Site, Vác
  - Research Site, Zalaegerszeg